CLINICAL TRIAL: NCT05211921
Title: A Single Arm Study to Confirm the Efficacy and Safety of Multi-Gyn ActiGel Plus for Treatment of Bacterial Vaginosis.
Brief Title: Single Arm Study of Multi-Gyn ActiGel Plus for Treatment of Bacterial Vaginosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karo Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21E3559
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-Gyn ActiGel Plus (Other): vaginal gel
  Interventions: Device: Multi-Gyn ActiGel Plus

INTERVENTIONS:
Device: Multi-Gyn ActiGel Plus — vaginal gel

SUMMARY:
Open, single arm trial that intends to confirm the safety and efficacy of Multi-Gyn ActiGel Plus for treatment of Bacterial Vaginosis. Adult women will be diagnosed by the gynaecologist based on the Amsel criteria at day 0. They will use the product for 7 days and will come to the practice at day 21. The primary endpoint is the clinical cure rate of Bacterial Vaginosis at 3 weeks after start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with BV (3 out of 4 Amsel criteria positive, with at least presence of clue cells (>20%)
* Women of childbearing potential
* Aged >18 years
* Signed written informed consent form
* Willing to comply to the follow-up schedule

Exclusion Criteria:

* Current clinically manifest of sexually transmitted gynecologically infection, genital tract infection, vulvovaginal candidosis or aerobic vaginitis
* Presence of Trichomonas and/or Candida Albicans in vaginal smear during examination of the smears for Amsel criteria (clue cells detection)
* Current genital malignancies
* Chemotherapy for any reason in last 6 months
* Radiotherapy in the genitourinary system in the last 12 months
* Use of antibiotics for any reason in the last 14 days
* Pregnancy or currently attempting to conceive
* Lactation
* Use of other treatment for vaginal conditions during the course of the clinical investigation
* Known allergies to ingredients of the product
* Concomitant medication for treatment of vaginal infections, or other use of intravaginal medication during the course of the clinical investigation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is clinical cure rate of BV at 3 weeks after start of treatment (Visit 2). | 3 weeks after start of treatment
  Primary endpoint is to demonstrate a responder rate significantly higher than 30% in treatment of bacterial vaginosis at 3 weeks after start of treatment using a two tailed binomial test.

SECONDARY OUTCOMES:
Relief of vaginal symptoms related to BV at Visit 2 | 3 weeks after start of treatment
  It is based on 0-10 point scale ( 0 is no improvement at all and 10 is the highest improvement)) . It is considered significant if the the score improvement is > 1.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Dermascan Poland, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No